CLINICAL TRIAL: NCT01792583
Title: The Nuvigil (Armodafinil) Tablets [C-IV]/Provigil (Modafinil) Tablets [C-IV] Pregnancy Registry
Brief Title: The Nuvigil and Provigil Pregnancy Registry
Status: Terminated | Type: Observational
Why Stopped: The study is no longer feasible.
Sponsor: Cephalon, Inc. (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Other Study IDs: C10953/9022
Record Dates: First submitted 2013-02-12; First posted 2013-02-15 (Estimated); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Narcolepsy; Obstructive Sleep Apnea; Shift Work Sleep Disorder
Keywords: pregnancy
MeSH Terms: conditions — Narcolepsy; Sleep Apnea, Obstructive; Sleep Disorders, Circadian Rhythm | interventions — Modafinil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 21 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Prospective Cohort: Prospective is defined per protocol: prospective data of pregnancy exposure are data acquired prior to the knowledge of the pregnancy outcome or prior to the detection of a congenital malformation at prenatal examination (e.g. fetal ultrasound, serum markers).
  Interventions: Drug: Modafinil/armodafinil
- Retrospective Cohort: Retrospective is defined per protocol: retrospective data of pregnancy exposure are data acquired after the outcome of the pregnancy is known or after the detection of a congenital malformation on prenatal examination.
  Interventions: Drug: Modafinil/armodafinil

INTERVENTIONS:
Drug: Modafinil/armodafinil
  Other Names: Provigil; Nuvigil

SUMMARY:
The primary objective of the Nuvigil/Provigil Pregnancy Registry is to characterize the pregnancy and fetal outcomes associated with Nuvigil and Provigil exposure during pregnancy.

DETAILED DESCRIPTION:
Both the prospective and the retrospective data are captured.

ELIGIBILITY:
Inclusion Criteria:

* Reported exposure to brand or generic formulations of Nuvigil (armodafinil) and/or Provigil (modafinil) within 6 weeks prior to becoming pregnant, or during pregnancy
* Patients who provide oral or written informed consent.
* Infant up to 1 year of age born to a female with maternal exposure to armodafinil and/or modafinil within 6 weeks prior to becoming pregnant or during pregnancy.
* Able and willing to provide healthcare professional and secondary contact information, and for the patient herself to be contacted periodically by Registry staff.

Exclusion Criteria:

* Patients who refuse to provide oral or written informed consent.
* Patients not exposed to armodafinil or modafinil within 6 weeks prior to becoming pregnant or during pregnancy.
* Infants whose mother was not exposed to armodafinil or modafinil within 6 weeks prior to becoming pregnant or during pregnancy.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The Registry is conducted in the US and includes female patients exposed to modafinil and/or armodafinil within 6 weeks prior to becoming pregnant or any time during pregnancy. The Registry is designed for open enrollment of all patients meeting the inclusion/exclusion criteria. Registry enrollment is initiated by either patients or healthcare professionals. Patients who meet the eligibility criteria and provide informed consent will be enrolled into the study.
Sampling Method: Non-Probability Sample
Enrollment: 191 (Actual)
Dates: Start 2009-06-30 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Incidence of major birth defects | End of pregnancy through the first year after delivery
  Major birth defects using Metropolitan Atlanta Congenital Birth Defects Program (MACDP) definitions

SECONDARY OUTCOMES:
Incidence of minor birth defects | End of pregnancy through the first year after delivery
Incidence of elective termination due to identified anomaly/birth defect or increased risk of anomaly/birth defect | Baseline and End of pregnancy
Incidence of spontaneous abortion (defined as <20 weeks gestation) | Baseline and End of pregnancy
Incidence of fetal death (defined as >=20 weeks gestation | Baseline and End of pregnancy
Incidence of neurodevelopmental problems | Baseline and End of pregnancy
Incidence of Microcephaly | End of pregnancy
Incidence of small size for gestational age | End of pregnancy
  defined as the observed weight of a live born infant or size of a fetus that is lower than expected on the basis of gestational age
Incidence of intrauterine growth restriction (IUGR) | End of pregnancy
  defined as observed fetal weight or birth weight below the 10th percentile for gestational age
Incidence of Low/very low birth weight (LBW/VLBW) | End of pregnancy
  Defines as - Low birth weight: <2500 g, regardless of gestational age and - Very low birth weight: birth weight <1500 g, regardless of gestational age
Incidence of Preterm delivery | End of pregnancy
Incidence of Preeclampsia/pregnancy-induced hypertension (PIH) | Baseline through End of pregnancy
Maternal breastmilk feeding practices | End of pregnancy through the first year after delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Teva Pregnancy Registry, West Chester, Pennsylvania, United States

REFERENCES:
- See also: Related Info — http://www.fda.gov/ScienceResearch/SpecialTopics/WomensHealthResearch/ucm134848.htm